CLINICAL TRIAL: NCT05892510
Title: Post-thrombectomy Intra-arterial Tenecteplase for Acute manaGement of Non-retrievable Thrombus and No-reflow in Emergent Stroke (EXTEND-AGNES TNK)
Brief Title: Post-thrombectomy Intra-arterial Tenecteplase for Acute manaGement of Non-retrievable Thrombus and No-reflow in Emergent Stroke
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT26024
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke, Acute; Cerebrovascular Disorders; Brain Disorder; Central Nervous System Diseases
Keywords: Tenecteplase; Fibrinolytic agents; Thrombectomy; No-reflow
MeSH Terms: conditions — Ischemic Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Intra-arterial bolus of placebo (0.9% Sodium Chloride solution) representing standard of care (no intra-arterial thrombolytic treatment).
  Interventions: Drug: Placebo
- Intra-arterial tenecteplase injection at the completion of thrombectomy (Experimental): intra-arterial tenecteplase (0.062mg/kg, maximum 6.25mg) administered as a bolus at the completion of thrombectomy through a microcatheter at the site of the initial-but-now-retrieved intracranial occlusion or in direct contact with the residual thrombus
  Interventions: Drug: Intra-arterial tenecteplase injection at the completion of thrombectomy

INTERVENTIONS:
Drug: Intra-arterial tenecteplase injection at the completion of thrombectomy — Intra-arterial tenecteplase (0.062mg/kg, maximum 6.25mg) administered as a bolus at the completion of thrombectomy through a microcatheter at the site of the initial-but-now-retrieved intracranial occlusion, or in direct contact with the residual thrombus
  Arms: Intra-arterial tenecteplase injection at the completion of thrombectomy
Drug: Placebo — intra-arterial bolus of 0.9% Sodium Chloride solution
  Arms: Placebo

SUMMARY:
Multicentre, prospective, Multi-arm Multi-stage (MAMS) seamless phase 2b/3 interventional randomized placebo-controlled double-blinded parallel-assignment (2 arms with 1:1 randomization) efficacy and safety trial to test intra-arterial tenecteplase at the completion of thrombectomy versus best practice in participants with anterior circulation LVO receiving mechanical thrombectomy within 24 hours of symptoms onset.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age≥18 years) presenting with ischemic stroke with arterial LVO on CT/MR Angiogram of the intracranial internal carotid or middle cerebral artery (MCA) first segment (M1) or proximal second segment (M2) committed to thrombectomy using standard criteria within 24 hours of onset:
* For 0-6 hours of symptom onset: Presence of arterial occlusion as defined above and ASPECTS≥3 on NCCT
* For 6-24 hours of symptom onset: Additional imaging criteria on CTP or MRI perfusion of core volume <100ml.
* Qualifying CT/MR within 4hrs of randomisation (repeat CT for transferred participants required if >4hr)
* Pre-stroke Modified Rankin Scale (mRS) score of ≤2 (mild pre-existing disability permitted)
* Local legal requirements for consent have been satisfied.

Exclusion Criteria:

* Intracranial hemorrhage identified by CT or MRI
* ASPECTS 0-2 on NCCT
* CTP or MRI perfusion ischemic core volume >100ml if presenting within 6-24 hours from symptoms onset
* Anticipated endovascular stenting required for intracranial or extracranial atherosclerotic stenosis/occlusion.
* More than six retrieval attempts in the same vessel
* Alteplase being infused within 30 minutes (~5x half-life) of anticipated trial drug administration
* Contraindication to imaging with contrast agents
* Any condition (eg.mid-arterial phase early venous filling) that in the judgment of investigators could impose hazards if study therapy is initiated
* Pregnant women.
* Current participation in another intervention research study that includes experimental interventions beyond standard-of-care.
* Anticoagulation. INR ≤1.7 if on warfarin, and dabigatran reversal by idarucizumab are permitted.
* Other standard contraindications to thrombolysis apart from time window.
* Known terminal illness such that the participants would not be expected to survive a year.
* Planned withdrawal of care or comfort care measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Early Neurological Improvement (Phase 2b) | 24-36 hours from time of randomisation
  Proportion of participants with Early Neurological Improvement (ENI) defined as NIHSS reduction>4
Functional independence (Phase 3) | 3 months
  Proportion of participants with Modified Rankin Scale (mRS) 0-2 (functional independence)

SECONDARY OUTCOMES:
Functional improvement | 3 months
  Reduction of ≥ 1 mRS category (ordinal analysis merging mRS categories 5-6)
Infarct growth | 24 hours
  Infarct growth volume on follow-up MRI or CT
No-reflow | 24 hours
  Proportion of participants with radiological no-reflow on MR perfusion or CTP
Symptomatic Intracerebral Hemorrhage | 36 hours
  Proportion of participants with sICH defined as parenchymal haematoma type 2 (PH2) or SAH/IVH within 36 hours combined with neurological deterioration leading to an increase of NIHSS ≥4 from baseline or leading to death
All cause mortality | 3 months
  Proportion of participants with death due to any cause
Quality of life assessment on EQ-5D | 3 months
  EQ-5D score

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (13):
  - Gold Coast Univeristy Hospital, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Royal Brisbane and Women's Hospital, Brisbane
  - Canberra Hospital, Canberra
  - Alfred Hospital, Melbourne
  - Austin Hospital, Melbourne
  - Monash Medical Centre, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - John Hunter Hospital, Newcastle
  - Fiona Stanley Hospital, Perth
  - Liverpool Hospital, Sydney
  - Royal North Shore Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No